CLINICAL TRIAL: NCT05138029
Title: Study on Precision Treatment of Diabetic Retinopathy Macular Edema Guided by Real-time Optical Coherence Tomography During Operation
Brief Title: Study on Precision Treatment of Diabetic Retinopathy Macular Edema Guided by Real-time OCT During Operation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MSZ20180
Record Dates: First submitted 2021-09-22; First posted 2021-11-30 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Ranibizumab; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Anti-VEGF treatment group (Experimental): Visual acuity and center thickness of the macula
  Interventions: Drug: Ranibizumab Injection [Lucentis]
- Inner limiting membrane stripping group (Experimental): Visual acuity and center thickness of the macula
  Interventions: Procedure: Inner limiting membrane stripping
- Glucocorticoid treatment group (Experimental): Visual acuity and center thickness of the macula
  Interventions: Drug: Dexamethasone intravitreal implant

INTERVENTIONS:
Drug: Ranibizumab Injection [Lucentis] — The visual acuity and the thickness of the center of the macula were reviewed at 1 day, 7 days, 1 month, 3 months, and 6 months after the operation to compare the effect of the operation, and observe the cornea, anterior chamber, vitreous cavity, and intraocular pressure.
  Other Names: Lucentis
  Arms: Anti-VEGF treatment group
Procedure: Inner limiting membrane stripping — The visual acuity and the thickness of the center of the macula were reviewed at 1 day, 7 days, 1 month, 3 months, and 6 months after the operation to compare the effect of the operation, and observe the cornea, anterior chamber, vitreous cavity, and intraocular pressure.
  Arms: Inner limiting membrane stripping group
Drug: Dexamethasone intravitreal implant — The visual acuity and the thickness of the center of the macula were reviewed at 1 day, 7 days, 1 month, 3 months, and 6 months after the operation to compare the effect of the operation, and observe the cornea, anterior chamber, vitreous cavity, and intraocular pressure.
  Other Names: Dexamethasone Implants
  Arms: Glucocorticoid treatment group

SUMMARY:
Select Proliferative Proliferative diabetic retinopathy(PDR) patients who are planning to undergo vitrectomy for informed notification. After obtaining informed consent, vitrectomy will be performed. After hemorrhage is removed, the macular shape can be obtained through intraoperative optical coherence tomography (iOCT) real-time scanning. If the central Macular Thickness (CMT) of the patient is ≥250μm, random Enter the Anti-vascular endothelial growth factor (anti-VEGF) treatment group, the internal limiting membrane stripping group and the glucocorticoid treatment group for treatment, and compare the patients' visual acuity (1 day, 7 days, 1 month, 3 months, 6 months) and The thickness of the center of the macula, compare and observe its treatment effect.

DETAILED DESCRIPTION:
1. Test method:

   * Include suitable cases of diabetic retinopathy and macular edema Inclusion criteria: a. PDR patients with severe vitreous hemorrhage who cannot collect oct images and require vitrectomy b. Type 2 diabetes, aged 18~80 years old c. Good blood sugar control (glycated hemoglobin <8.3%) d. Sign the informed consent form voluntarily, and are willing and able to follow the outpatient visits and research procedures within the time specified in the trial Exclusion criteria: a. Exclude severe infections of conjunctiva, cornea, and sclera b. Combined with other retinal vascular diseases such as retinal vein occlusion c. Cardiorenal insufficiency d. Myocardial infarction or stroke occurred within 6 months ②Intraoperative real-time operation All patients underwent 25Gauge(25G) transplanter three-channel vitrectomy to remove cloudy vitreous or vitreous hemorrhage and posterior vitreous cortex. Through intraoperative oct, the macular area was observed in real time and the central macular thickness was measured. If central macular thickness (CMT) ≥ 250 μm, anti-VEGF, glucocorticoid, or internal limiting membrane peeling was randomly selected to treat macular edema.

     * Re-examine the effect of surgery after operation The visual acuity and the thickness of the center of the macula were reviewed at 1 day, 7 days, 1 month, 3 months, and 6 months after the operation to compare the effect of the operation, and observe the cornea, anterior chamber, vitreous cavity, and intraocular pressure.

ELIGIBILITY:
Inclusion Criteria:

* PDR patients with severe vitreous hemorrhage who cannot collect oct images and need vitrectomy
* Type 2 diabetes, aged 18~80 years old
* Good blood sugar control (glycated hemoglobin <8.3%)
* Sign the informed consent form voluntarily, and are willing and able to follow the outpatient visits and research procedures within the time specified in the trial

Exclusion Criteria:

* Exclude severe infections of conjunctiva, cornea, and sclera
* Combined with other retinal vascular diseases such as retinal vein occlusion
* Cardiorenal insufficiency
* Myocardial infarction or stroke occurred within 6 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-11-15 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Review the patient's vision before surgery | The day before the patient's surgery
  Optical Coherence Tomography (OCT) is currently the main examination method for measuring retinal thickness and evaluating DME morphology and fine structure. DME OCT examination has a variety of morphological manifestations and accompanying images, and various manifestations reflect different pathological basis.

SECONDARY OUTCOMES:
Review the patient's vision for one day after surgery | The patient's first day after surgery
  Optical Coherence Tomography (OCT) is currently the main examination method for measuring retinal thickness and evaluating DME morphology and fine structure. DME OCT examination has a variety of morphological manifestations and accompanying images, and various manifestations reflect different pathological basis.
Review the patient's vision for 7 days after surgery | 1st week after surgery
  Optical Coherence Tomography (OCT) is currently the main examination method for measuring retinal thickness and evaluating DME morphology and fine structure. DME OCT examination has a variety of morphological manifestations and accompanying images, and various manifestations reflect different pathological basis.
Review the patient's vision for 1 month after surgery | 4th week after surgery
  Optical Coherence Tomography (OCT) is currently the main examination method for measuring retinal thickness and evaluating DME morphology and fine structure. DME OCT examination has a variety of morphological manifestations and accompanying images, and various manifestations reflect different pathological basis.
Review the patient's vision for 3 months after surgery | 12th week after surgery
  Optical Coherence Tomography (OCT) is currently the main examination method for measuring retinal thickness and evaluating DME morphology and fine structure. DME OCT examination has a variety of morphological manifestations and accompanying images, and various manifestations reflect different pathological basis.
Review the patient's vision for 6 months after surgery | 24th week after surgery
  Optical Coherence Tomography (OCT) is currently the main examination method for measuring retinal thickness and evaluating DME morphology and fine structure. DME OCT examination has a variety of morphological manifestations and accompanying images, and various manifestations reflect different pathological basis.

CONTACTS AND LOCATIONS:
Overall Officials: Rongrong Zhu, master, Principal Investigator — Affiliated Hospital of Nantong University
Locations (1):
- Affiliated Hospital of Nantong University, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No